CLINICAL TRIAL: NCT05849753
Title: Breaking Health Care Disparities in Access to Advanced Diabetes Technologies in Children With Type 1 Diabetes
Brief Title: Breaking Disparities in Access to Advanced Diabetes Technologies in Children With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Principal Investigator, Nelly Mauras, Vice Chair of Pediatrics for Research/Director of Research, Nemours North FL, Nemours Children's Clinic
Other Study IDs: 1980589-3]
Record Dates: First submitted 2023-03-26; First posted 2023-05-09 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 1; Child; Delivery of Health Care; Equipment and Supplies
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- T1DM lower SES: Type 1 diabetes of lower SES, including AA and Latino racial/ethnic minorities, who are in suboptimal diabetes control.
  Interventions: Device: Advanced artificial pancreas closed-loop technology

INTERVENTIONS:
Device: Advanced artificial pancreas closed-loop technology — Study is an observational capture of data in patients that qualify, before and after the use of any FDA-approved closed-loop system of Subject's/Family's choosing that uses a CGM that does not require fingerprick calibrations. Devices prescribed available through their insurance (including Medicaid).

SUMMARY:
50 children/adolescents (ages 6 to <18yrs) with T1D in suboptimal control (HbA1c≥8.0%) and lower SES (below 200% poverty line) on insulin therapy (either injections or open-loop pumps) will be recruited at Nemours ~ 1/3 each AA, Hispanic/Latino, non-Hispanic whites. All families that qualify and agree to transition to closed-loop technologies will be recruited to allow data to be gathered before and after use of devices. They will go through the process of approval with the assistance of an insurance navigator in clinic. Those not a CGM will be prescribed one as well. Diabetes care will be 'real life', devices will be prescribed, and care per clinic routine with periodic device downloads. Principal outcome, time-in-range, will be analyzed at 3-months compared to baseline, each participant their own control. Secondary outcomes including HbA1c, other glucose metrics and questionnaires related to use of technology and diabetes distress will be also analyzed. All outcomes will also be collected at 6-months. Results could have important and fast applicability to the field and help better inform decision makers, including payers, clinicians, and patients and families and could serve to decrease health care disparities in this needy population.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) has serious complications, yet only ~17% of children achieve an HbA1C goal of <7.5% and in adolescents mean HbA1c remains persistently high at 9.3%. Technology use in children has increased, both insulin pump use and continuous glucose monitors (CGM), offering hope to improve diabetes control and outcomes. There are however, striking socio-economic (SES) and racial/ethnic disparities in these outcomes, with worse metabolic control and much lower use of technology in those of lower SES and racial/ethnic minorities. Reasons are multifactorial, including more limited access to care, insurance challenges, and providers' biases in prescribing these devices, but also related to implicit bias and structural racism towards minority groups. Rates of diabetes complications and ketoacidosis are higher in Black and Latino youth, yet these children are largely under-represented in clinical trials and in the clinical use of FDA-approved modern diabetes technologies. Closed-loop artificial pancreas now allows for the semi-automatic or fully automatic delivery of insulin based on CGM glucose, with potential to further improve glycemic control. The investigators' recent data suggest that patients in ethnic minority groups provided devices through a clinical trial may indeed benefit from this technology with improved time-in-range and HbA1c. Insurance companies, including Medicaid now include these FDA-approved devices in their formulary, yet they continue to be underutilized by these needy families. The investigators believe the overwhelming amount of data support the routine use of closed-loop insulin delivery technology in children. The proposed study will be first to compare use of advanced closed-loop insulin delivery systems specifically focused on children with T1D of lower SES, including racial/ethnic minorities, using patient-centered outcomes while understanding clinical markers of diabetic control. The principal study question is whether these children can benefit from a closed-loop insulin delivery treatment option and improve health care disparities in a 'real life' setting.

Specific Aims:

To investigate in children with type 1 diabetes of lower SES, including AA and Latino racial/ethnic minorities, who are in suboptimal diabetes control, if when they are consistently offered advanced artificial pancreas closed-loop technology, and are better assisted in getting approval and starting these devices clinically:

1. can health care disparities decrease by improving overall diabetes control including time-in-range sensor glucose(70-180mg/dl) (principal) and other metrics of glycemic control including HbA1c at 3 months;
2. can any clinical benefit be sustained for 6 months in a real life setting;
3. can the above treatments improve patient/family reported perceptions of quality of life, including diabetes distress and psychosocial aspects of closed-loop technology? (secondary)

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of T1D for at least 1 year based on clinical presentation (polyuria, polydipsia, weight loss, and/or ketoacidosis, or with positive diabetes autoantibodies) on insulin, including injections or open-loop pumps

* HbA1C ≥ 8.0% at least twice within the last 12 months before study initiation, upper limit of HbA1C <14%
* Be of lower SES, defined based on < 200% above published US levels of poverty by family size and income, or based on exceptional circumstantial needs in the opinion of the investigators
* Approximately 1/3 AA, 1/3 Hispanic/Latinos, 1/3 non-Hispanic whites. Asians, Pacific Islanders and other ethnic groups however will not be excluded from participation if other criteria met
* History of hypothyroidism on adequate replacement therapy with normal thyroid function will be allowed

Exclusion Criteria:

* Severe eczema or any other skin condition that would limit availability of healthy skin to wear devices
* Chronic medications/medical conditions that could interfere with diabetes management (ADHD medications allowed)
* Chronic seizures, or severe neurodevelopmental delay
* Current use of hybrid closed-loop, automated insulin delivery system
* Significant mental health disorder that in opinion of the investigator would hinder device use

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A target of 50 children and adolescents (ages 6 to <18yrs) with T1D in suboptimal control (HbA1c≥8.0%) and of lower SES (below 200% of state-specific poverty line by family size and income), with no other chronic illnesses will be recruited from the Pediatric Endocrine clinics at Nemours Children's Health Clinics in Jacksonville and Orlando, FL. Cohort will be ~ 1/3 each AA, Hispanic/Latino, and non-Hispanic White (NHW).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Percent sensor glucose time-in-range | 3 months
  70-180mg/dL

SECONDARY OUTCOMES:
HbA1C | 3 months
  percent
Percent sensor glucose time in hypoglycemic range | 3 months
  less than 54 mg/dL
Perceptions of Benefits & Burden of Closed-Loop Systems | 3 months
  Psychosocial questionnaire (Scale: 35-175); higher score reflects better outcome
Problem Areas in Diabetes | 3 months
  Psychosocial questionnaire (Scale: 0-80); lower score reflects better outcome
Technology Attitudes | 3 months
  Psychosocial questionnaire related to diabetes technology (Scale: 5-25); higher score reflects better outcome
Percent sensor glucose time-in-range | 6 months
  70-180mg/dL
HbA1C | 6 months
  percent
Percent sensor glucose time in hypoglycemic range | 6 months
  less than 54 mg/dL
Perceptions of Benefits & Burden of Closed-Loop Systems | 6 months
  Psychosocial questionnaire (Scale: 35-175); higher score reflects better outcome
Problem Areas in Diabetes | 6 months
  Psychosocial questionnaire (Scale: 0-80); lower score reflects better outcome
Technology Attitudes | 6 months
  Psychosocial questionnaire relating to diabetes technology (Scale: 5-25); higher score reflects better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Health Jacksonville
Locations (2):
- United States (2):
  - Nemours Children's Health, Jacksonville, Florida
  - Nemours Children's Health, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided